CLINICAL TRIAL: NCT06952504
Title: A Phase 3 Randomized, Open-label, Multicenter Study to Compare the Efficacy and Safety of Sacituzumab Tirumotecan (Sac-TMT, MK-2870) in Combination With Pembrolizumab Versus Pembrolizumab Alone as First-line Maintenance Treatment in Participants With Mismatch Repair Proficient Endometrial Cancer (TroFuse-033/GOG-3119/ENGOT-en29)
Brief Title: A Study to Compare Sacituzumab Tirumotecan (MK-2870) in Combination With Pembrolizumab (MK-3475) Versus Pembrolizumab Alone as Treatment in Participants With Mismatch Repair Proficient Endometrial Cancer (MK-2870-033/TroFuse-033/GOG-3119/ENGOT-en29)
Acronym: TroFuse-033
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2870-033; 2024-519331-42-00 (Registry Identifier: EU CT); U1111-1315-0794 (Registry Identifier: UTN); GOG-3119 (Other: Gynecologic Oncology Group); ENGOT-en29 (Other: European Network for Gynaecological Oncological Trial groups); TroFuse-033 (Other: MSD); jRCT2011250020 (Registry Identifier: Japan Registry of Clinical Trial (jRCT))
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Trophoblast cell surface antigen 2 (TROP2)
MeSH Terms: conditions — Endometrial Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Paclitaxel; Docetaxel

STUDY DESIGN:
Intervention Model Description: Participants are allocated to a single induction arm, then assigned randomly to either one of two maintenance treatment arms or one of two subsequent treatment arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Maintenance Treatment Arm A: Pembrolizumab + Sacituzumab Tirumotecan (Experimental): During the Induction Phase, participants receive pembrolizumab 200 mg, carboplatin area under the curve (AUC) 5 (mg/mL/min), and paclitaxel 175 mg/m2 or docetaxel 75 mg/m2 on Day 1 of each 3-week cycle for 6 cycles (up to approximately 4 months).
  During the Maintenance Treatment Phase, participants receive sac-TMT 4 mg/kg on Days 1, 15, and 29 of each 6-week cycle and pembrolizumab 400 mg on Day 1 of each 6-week cycle for up to 14 cycles (up to approximately 19 months).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Docetaxel; Biological: Sacituzumab Tirumotecan
- Maintenance Treatment Arm B: Pembrolizumab Monotherapy (Active Comparator): During the Induction Phase, participants receive pembrolizumab 200 mg, carboplatin AUC 5 (mg/mL/min), and paclitaxel 175 mg/m2 or docetaxel 75 mg/m2 on Day 1 of each 3-week cycle for 6 cycles (up to approximately 4 months).
  During the Maintenance Treatment Phase, participants receive pembrolizumab 400 mg on Day 1 of each 6-week cycle for up to 14 cycles (up to approximately 19 months).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Docetaxel
- Subsequent Treatment Arm A: Pembrolizumab + Sacituzumab Tirumotecan (Experimental): During the Induction Phase, participants receive pembrolizumab 200 mg, carboplatin AUC 5 (mg/mL/min), and paclitaxel 175 mg/m2 or docetaxel 75 mg/m2 on Day 1 of each 3-week cycle for 6 cycles (up to approximately 4 months).
  During the Subsequent Treatment Phase, participants receive sac-TMT 4 mg/kg on Days 1, 15, and 29 of each 6-week cycle until discontinuation criteria is met and pembrolizumab 400 mg on Day 1 of each 6-week cycle for up to 14 cycles (up to approximately 19 months).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Docetaxel; Biological: Sacituzumab Tirumotecan
- Subsequent Treatment Arm B: Sacituzumab Tirumotecan Monotherapy (Active Comparator): During the Induction Phase, participants receive pembrolizumab 200 mg, carboplatin AUC 5 (mg/mL/min), and paclitaxel 175 mg/m2 or docetaxel 75 mg/m2 on Day 1 of each 3-week cycle for 6 cycles (up to approximately 4 months).
  During the Subsequent Treatment Phase, participants receive sac-TMT 4 mg/kg on Days 1, 15, and 29 of each 6-week cycle until discontinuation criteria is met.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Docetaxel; Biological: Sacituzumab Tirumotecan

INTERVENTIONS:
Biological: Pembrolizumab — Intravenous (IV) Infusion
  Other Names: KEYTRUDA®; MK-3475; SCH 900475
  Arms: Maintenance Treatment Arm A: Pembrolizumab + Sacituzumab Tirumotecan; Maintenance Treatment Arm B: Pembrolizumab Monotherapy; Subsequent Treatment Arm A: Pembrolizumab + Sacituzumab Tirumotecan
Drug: Carboplatin — During the Induction Phase, participants receive carboplatin AUC 5 (mg/mL/min) on Day 1 of each 3-week cycle for 6 cycles (up to approximately 4 months) via IV infusion.
Drug: Paclitaxel — During the Induction Phase, participants receive paclitaxel 175 mg/m2 on Day 1 of each 3-week cycle for 6 cycles (up to approximately 4 months) via IV infusion.
Drug: Docetaxel — During the Induction Phase, participants may receive docetaxel (in place of paclitaxel) 75 mg/m2 on Day 1 of each 3-week cycle for 6 cycles (up to approximately 4 months) via IV infusion.
Biological: Sacituzumab Tirumotecan — IV Infusion
  Other Names: sac-TMT; MK-2870; SKB264
  Arms: Maintenance Treatment Arm A: Pembrolizumab + Sacituzumab Tirumotecan; Subsequent Treatment Arm A: Pembrolizumab + Sacituzumab Tirumotecan; Subsequent Treatment Arm B: Sacituzumab Tirumotecan Monotherapy

SUMMARY:
Researchers are looking for new ways to treat people with proficient mismatch repair (pMMR) endometrial cancer (EC) that is advanced or recurrent.

* EC is a type of cancer that starts in the tissues inside the uterus (womb)
* pMMR indicates that certain normal proteins are present in the cancer cells
* Advanced means the cancer has spread locally or to other parts of the body (metastatic) and cannot be removed with surgery
* Recurrent means the cancer came back after surgery

Sacituzumab tirumotecan (also known as sac-TMT) and pembrolizumab are the study medicines. Sac-TMT is an antibody drug conjugate (ADC). An ADC attaches to specific targets on cancer cells and delivers treatment to destroy those cells.

The goal of this study is to learn if people who receive sac-TMT with pembrolizumab live longer and without the cancer getting worse compared to people who receive pembrolizumab alone.

DETAILED DESCRIPTION:
All participants undergo an initial Induction Phase of six cycles, each cycle consisting of pembrolizumab + carboplatin + paclitaxel or docetaxel. Each cycle is three weeks. Participants whose cancer does not progress enter the Maintenance Treatment Phase and are then randomly assigned to pembrolizumab + sac-TMT or pembrolizumab monotherapy. Participants whose cancer does progress will have the possibility to enter the Subsequent Treatment Phase and are then randomly assigned to pembrolizumab + sac-TMT or sac-TMT monotherapy.

ELIGIBILITY:
Key inclusion criteria include but are not limited to:

* Has a histologically confirmed diagnosis of primary advanced or recurrent endometrial carcinoma that has been confirmed as proficient mismatch repair (pMMR)
* Has radiographically evaluable disease, with measurable Stage III or either measurable or non-measurable Stage IV or recurrent disease per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1), as assessed by the investigator.
* Has received no prior systemic therapy for endometrial carcinoma except the following conditions as pre-specified by the protocol: 1 prior line of systemic platinum-based adjuvant and/or neoadjuvant chemotherapy in the setting of curative-intent, prior radiation with or without radiosensitizing chemotherapy if >2 weeks before the start of induction treatment, or prior hormonal therapy for treatment of endometrial carcinoma that was discontinued ≥1 week before the start of induction treatment

Key exclusion criteria include but are not limited to:

* Has carcinosarcoma, neuroendocrine tumors or endometrial sarcoma, including stromal sarcoma, leiomyosarcoma, adenosarcoma, or other types of sarcomas
* Has endometrial carcinoma of any histology that is mismatch repair deficient (dMMR)
* Is a candidate for curative-intent surgery or curative-intent radiotherapy at the time of enrollment
* Has a history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Human Immunodeficiency Virus-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Received prior therapy in any setting with any of the following: anti-programmed cell death 1 protein, anti-programmed cell death ligand 1, anti-programmed cell death ligand 2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor; trophoblast cell surface antigen 2-targeted antibody drug conjugate; or topoisomerase I inhibitor-containing antibody drug conjugate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1123 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2032-05-24 (Estimated); Study Completion 2032-05-24 (Estimated)

PRIMARY OUTCOMES:
Maintenance Treatment: Progression-Free Survival (PFS) | Up to approximately 44 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as evaluated by the blinded independent central review (BICR). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Maintenance Treatment: Overall Survival (OS) | Up to approximately 54 months
  OS is defined as time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Maintenance Treatment: Progression-Free Survival 2 (PFS2) as Assessed by Investigator | Up to approximately 54 months
  PFS2 is defined as the time from randomization to the documented subsequent objective disease progression after initiation of new anticancer therapy or death due to any cause, whichever occurs first. PFS2 as assessed by the investigator will be presented.
Maintenance Treatment: Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 27 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Maintenance Treatment: Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Maintenance Treatment: Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Item Mean Score | Baseline and up to approximately 24 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7- point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 mean score will be presented.
Maintenance Treatment: Change from baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) Combined Score | Baseline and up to approximately 24 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life of cancer patients. The physical functioning score is based on participant responses to questions scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate better physical functioning. The change from baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) combined score will be presented.
Maintenance Treatment: Change from baseline in EORTC QLQ-C30 Role Functioning (Items 6 and 7) Combined Score | Baseline and up to approximately 24 months
  EORTC QLQ-C30 is a 30-item scale to assess the overall quality of life of cancer patients. The role functioning score is based on participant responses to questions scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate better role functioning. The change from baseline in EORTC QLQ-C30 Role Functioning (Items 6 and 7) combined score will be presented.
Maintenance Treatment: Change from baseline in EORTC QLQ Endometrial Cancer Symptom Score (QLQ-EN24) | Baseline and up to approximately 24 months
  The EORTC-QLQ-EN24 is a 24-item questionnaire developed to be used in conjunction with the EORTC-QLQ-C30 to assess the quality of life of endometrial cancer patients. Participant responses are scored on a 4-point scale (1=not at all to 4=very much). A higher score indicates a better quality of life. The change from baseline in EORTC QLQ-E24 back and pelvis pain score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (220):
- United States (36):
  - University of South Alabama, Mitchell Cancer Institute ( Site 6033), Mobile, Alabama
  - Alaska Women's Cancer Care ( Site 6036), Anchorage, Alaska
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 6020), Orange, California
  - Yale University School of Medicine ( Site 6009), New Haven, Connecticut
  - MedStar Washington Hospital Center ( Site 5005), Washington D.C., District of Columbia
  - Florida Cancer Specialists - South ( Site 7003), Fort Myers, Florida
  - UF Health Davis Cancer Pavilion and Shands Med Plaza ( Site 6026), Gainesville, Florida
  - Mount Sinai Cancer Center ( Site 6031), Miami Beach, Florida
  - Florida Cancer Specialists ( Site 7002), St. Petersburg, Florida
  - Florida Cancer Specialists East ( Site 7001), West Palm Beach, Florida
  - St. Joseph's/Candler Health System ( Site 6021), Savannah, Georgia
  - University of Chicago Medical Center ( Site 5002), Chicago, Illinois
  - Parkview Research Center ( Site 6008), Fort Wayne, Indiana
  - Women's Cancer Care ( Site 6010), Covington, Louisiana
  - TRIALS 365 ( Site 6005), Shreveport, Louisiana
  - Maine Medical Center - Scarborough Campus ( Site 6042), Scarborough, Maine
  - Minnesota Oncology Hematology, PA ( Site 8003), Minneapolis, Minnesota
  - St. Dominic's Hospital ( Site 5004), Jackson, Mississippi
  - Holy Name Medical Center ( Site 6011), Teaneck, New Jersey
  - University of New Mexico Comprehensive Cancer Center ( Site 6046), Albuquerque, New Mexico
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 6055), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone ( Site 6004), New York, New York
  - Duke Cancer Institute ( Site 6049), Durham, North Carolina
  - FirstHealth of the Carolinas ( Site 6037), Pinehurst, North Carolina
  - Miami Valley Hospital South ( Site 6014), Centerville, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 6047), Tulsa, Oklahoma
  - St. Luke's University Health Network ( Site 6041), Bethlehem, Pennsylvania
  - Hospital of the University of Pennsylvania ( Site 5007), Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania ( Site 6023), Philadelphia, Pennsylvania
  - AHN West Penn Hospital ( Site 6006), Pittsburgh, Pennsylvania
  - Women & Infants Hospital ( Site 5003), Providence, Rhode Island
  - Texas Oncology - DFW ( Site 8004), Fort Worth, Texas
  - Texas Oncology-San Antonio Medical Center ( Site 8001), San Antonio, Texas
  - Texas Oncology - Northeast Texas ( Site 8002), Tyler, Texas
  - Inova Schar Cancer Institute ( Site 6003), Fairfax, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 5000), Richmond, Virginia
- Argentina (5):
  - Instituto Alexander Fleming ( Site 0105), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0108), Mar del Plata, Buenos Aires
  - Fundación Respirar ( Site 0101), Buenos Aires, Buenos Aires F.D.
  - Hospital Británico de Buenos Aires ( Site 0103), CABA
  - Instituto San Marcos ( Site 0106), San Juan
- Australia (3):
  - Blacktown Hospital ( Site 0201), Blacktown, New South Wales
  - Royal Brisbane and Women's Hospital ( Site 0206), Brisbane, Queensland
  - Epworth Freemasons ( Site 0207), Melbourne, Victoria
- Austria (3):
  - Medizinische Universität Graz-Abteilung für Gynäkologie / Onkologie ( Site 0303), Graz, Styria
  - Medizinische Universitaet Innsbruck-Univ.-Klinik f. Gynäkologie und Geburtshilfe ( Site 0301), Innsbruck, Tyrol
  - Medizinische Universität Wien - Allg. Gynaekologie & Gyn. Onkologie ( Site 0302), Vienna
- Belgium (5):
  - CHU Saint-Pierre ( Site 0405), Brussels, Bruxelles-Capitale, Region de
  - AZ Maria Middelares ( Site 0402), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0401), Leuven, Vlaams-Brabant
  - Grand Hôpital de Charleroi ( Site 0403), Charleroi, Wallonne, Region
  - CHU de Liege ( Site 0404), Liège, Wallonne, Region
- Brazil (4):
  - Hospital Araújo Jorge ( Site 0521), Goiânia, Goiás
  - Hospital São Lucas da PUCRS ( Site 0522), Porto Alegre, Rio Grande do Sul
  - IBCC - Instituto Brasileiro de Controle do Câncer ( Site 0525), São Paulo, São Paulo
  - Instituto Nacional de Câncer - INCA ( Site 0515), Rio de Janeiro
- Canada (8):
  - CancerCare Manitoba ( Site 0617), Winnipeg, Manitoba
  - Sault Area Hospital ( Site 0616), Sault Ste. Marie, Ontario
  - Sunnybrook Research Institute ( Site 0610), Toronto, Ontario
  - Princess Margaret Cancer Center ( Site 0609), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0605), Montreal, Quebec
  - Jewish General Hospital ( Site 0606), Montreal, Quebec
  - McGill University Health Centre ( Site 0604), Montreal, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0608), Sherbrooke, Quebec
- Chile (5):
  - Centro de Estudios Clínicos SAGA ( Site 0708), Santiago, Region M. de Santiago
  - FALP ( Site 0702), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0705), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0703), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS ( Site 0704), Viña del Mar, Región de Valparaíso
- China (29):
  - Peking University Peoples Hospital ( Site 0845), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 0838), Chongqing, Chongqing Municipality
  - Fujian Province Cancer Hospital ( Site 0802), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 0822), Xiamen, Fujian
  - Sun Yat-sen University Cancer Center ( Site 0846), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University ( Site 0801), Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University ( Site 0829), Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College ( Site 0827), Shantou, Guangdong
  - Affiliated Hospital of Guangdong Medical University ( Site 0823), Zhanjiang, Guangdong
  - Liuzhou People's Hospital ( Site 0831), Liuchow, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital. ( Site 0825), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital ( Site 0850), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0806), Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University ( Site 0833), Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center ( Site 0824), Wuhan, Hubei
  - Xiangya Hospital Central South University ( Site 0821), Changsha, Hunan
  - Nanjing First Hospital ( Site 0828), Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital ( Site 0807), Nanchang, Jiangxi
  - The First Hospital Of Jilin University ( Site 0815), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 0816), Xi'an, Shaanxi
  - Shandong Cancer Hospital ( Site 0803), Jinan, Shandong
  - Shanghai Tenth People's Hospital ( Site 0847), Shanghai, Shanghai Municipality
  - Obstetrics & Gynecology Hospital of Fudan University ( Site 0818), Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital ( Site 0843), Taiyuan, Shanxi
  - The Second People's Hospital of Yibin ( Site 0840), Yibin, Sichuan
  - Yunnan Province Cancer Hospital ( Site 0811), Kunming, Yunnan
  - The Affiliated Women's Hospital of Zhejiang University ( Site 0834), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 0809), Linhai, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 0805), Wenzhou, Zhejiang
- Colombia (4):
  - Instituto de Cancerología S.A.S ( Site 0904), Medellín, Antioquia
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 0905), Medellín, Antioquia
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0902), Bogotá, Bogota D.C.
  - Oncologos Del Occidente ( Site 0907), Pereira, Risaralda Department
- Czechia (4):
  - Fakultni nemocnice Ostrava ( Site 1104), Ostrava, Ostrava Mesto
  - Nemocnice AGEL Novy Jicin a.s. ( Site 1102), Nový Jičín
  - Vseobecna fakultni nemocnice v Praze-Gynekologicko-porodnicka klinika 1.LF a VFN ( Site 1101), Prague
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 1103), Prague
- Denmark (4):
  - Herlev and Gentofte Hospital ( Site 1202), Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby ( Site 1205), Aarhus, Central Jutland
  - Aalborg Universitetshospital, Syd ( Site 1203), Aalborg, North Denmark
  - Roskilde Sygehus ( Site 1204), Roskilde, Region Sjælland
- Finland (4):
  - Kuopion Yliopistollinen Sairaala ( Site 1304), Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala ( Site 1303), Tampere, Pirkanmaa
  - Turku University Hospital-Department of Obstetrics and Gynecology ( Site 1302), Turku, Southwest Finland
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 1301), Helsinki, Uusimaa
- France (10):
  - Institut Paoli Calmettes ( Site 1410), Marseille, Bouches-du-Rhone
  - Centre Francois Baclesse ( Site 1412), Caen, Calvados
  - Hôpital Privé Des Côtes d'Armor ( Site 1404), Plérin, Cotes-d Armor
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest ( Site 1405), Bordeaux, Gironde
  - Oncopole Claudius Regaud ( Site 1407), Toulouse, Haute-Garonne
  - Institut Curie - site Saint-Cloud ( Site 1408), Saint-Cloud, Hauts-de-Seine
  - Institut De Cancerologie De L Ouest ( Site 1403), Saint-Herblain, Loire-Atlantique
  - CENTRE LEON BERARD ( Site 1401), Lyon, Rhone
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 1411), Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon ( Site 1409), Paris
- Germany (5):
  - Klinikum Mutterhaus der Borromäerinnen ( Site 1506), Trier, Rhineland-Palatinate
  - CaritasKlinikum Saarbruecken St. Theresia ( Site 1508), Saarbrücken, Saarland
  - Universitaetsklinikum Jena ( Site 1503), Jena, Thuringia
  - Charité Campus Virchow-Klinikum ( Site 1501), Berlin
  - Asklepios Kliniken Hamburg ( Site 1509), Hamburg
- Greece (5):
  - Alexandra General Hospital of Athens ( Site 1604), Athens, Attica
  - Aretaieio Hospital ( Site 1602), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL ( Site 1603), Chaïdári, Attica
  - Iaso Genera ( Site 1605), Marousi, Attica
  - Agios Loukas Clinic-DEPARTMENT OF ONCOLOGY ( Site 1601), Thessaloniki, Central Macedonia
- Debreceni Egyetem Klinikai Kozpont-Szülészeti és Nőgyógyászati Klinika ( Site 1701), Debrecen, Hungary
- Ireland (2):
  - Mater Misericordiae University Hospital ( Site 1904), Dublin
  - St. James's Hospital ( Site 1901), Dublin
- Israel (5):
  - Rambam Health Care Campus ( Site 2025), Haifa
  - Carmel Hospital ( Site 2023), Haifa
  - Shaare Zedek Medical Center ( Site 2020), Jerusalem
  - Meir Medical Center. ( Site 2021), Kfar Saba
  - Sourasky Medical Center ( Site 2022), Tel Aviv
- Italy (13):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori" ( Site 2107), Meldola, Forli-Cesena
  - Ospedale Humanitas San Pio X ( Site 2106), Milan, Lombardy
  - Ospedale Cannizzaro ( Site 2103), Catania
  - Azienda Ospedaliera Universitaria Careggi ( Site 2109), Florence
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 2114), Milan
  - Istituto Europeo di Oncologia ( Site 2110), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 2104), Napoli
  - Azienda Ospedaliero Universitaria Pisana Ospedale S. Chiara ( Site 2108), Pisa
  - Istituto Nazionale Tumori Regina Elena ( Site 2102), Roma
  - Fondazione Policlinico Universitario Agostino Gemelli ( Site 2105), Roma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino ( Site 2111), Torino
  - Ospedale Mauriziano ( Site 2101), Torino
  - Ospedale Santa Maria di Ca' Foncello ( Site 2112), Treviso
- Japan (14):
  - National Hospital Organization Shikoku Cancer Center ( Site 2206), Matsuyama, Ehime
  - Ehime University Hospital ( Site 2213), Tōon, Ehime
  - Kurume University Hospital ( Site 2204), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 2202), Ōta, Gunma
  - National Hospital Organization Hokkaido Cancer Center ( Site 2212), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 2216), Akashi, Hyōgo
  - Iwate Medical University Hospital ( Site 2207), Shiwa-gun, Iwate
  - Saitama Medical University International Medical Center ( Site 2201), Hidaka, Saitama
  - National Cancer Center Hospital ( Site 2211), Chūō, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 2208), Koto, Tokyo
  - Keio University Hospital ( Site 2209), Shinjuku, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 2203), Fukuoka
  - Niigata Cancer Center Hospital ( Site 2210), Niigata
  - Okayama University Hospital ( Site 2215), Okayama
- Maastricht UMC+ ( Site 2501), Maastricht, Limburg, Netherlands
- Norway (3):
  - Stavanger Universitetssykehus ( Site 2703), Norway, Rogaland
  - Universitetssykehuset Nord-Norge HF ( Site 2702), Tromsø, Troms
  - Oslo universitetssykehus, Radiumhospitalet ( Site 2701), Oslo
- Peru (3):
  - Clínica San Felipe ( Site 2804), Jesus Maria, Lima region
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 2803), San Isidro, Lima region
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS ( Site 2805), Lima
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 3011), Poznan, Greater Poland Voivodeship
  - Wielkopolskie Centrum Onkologii im. Marii Skłodowskiej-Curie ( Site 3003), Poznan, Greater Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 3004), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 3002), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Ginekologii, Ginekologii Onkologicznej i Endokrynologii Gi ( Site 3001), Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 3006), Gliwice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii. ( Site 3008), Kielce, Świętokrzyskie Voivodeship
- Puerto Rico Cancer Specialists Clinical Trials ( Site 4201), San Juan, Puerto Rico
- Singapore (2):
  - National University Hospital ( Site 3202), Singapore, Central Singapore
  - National Cancer Centre Singapore ( Site 3201), Singapore, Central Singapore
- South Korea (6):
  - National Cancer Center ( Site 3106), Gyeonggi-do, Kyonggi-do
  - Keimyung University Dongsan Hospital ( Site 3105), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 3102), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 3101), Seoul
  - Asan Medical Center ( Site 3103), Seoul
  - Samsung Medical Center ( Site 3104), Seoul
- Spain (7):
  - Institut Català d'Oncologia - L'Hospitalet ( Site 3408), L'Hospitalet de Llobregat, Barcelona
  - Institut Català d'Oncologia (ICO) - Girona ( Site 3407), Girona, Gerona
  - Hospital Universitari Vall d''Hebron ( Site 3401), Barcelona
  - Hospital Universitario Reina Sofia ( Site 3402), Córdoba
  - Hospital Universitario Ramon y Cajal ( Site 3403), Madrid
  - Hospital Universitario 12 de Octubre ( Site 3404), Madrid
  - Fundación Instituto Valenciano de Oncología ( Site 3405), Valencia
- Sweden (2):
  - Skånes Universitetssjukhus Lund ( Site 3502), Lund, Skåne County
  - Akademiska Sjukhuset ( Site 3501), Uppsala, Uppsala County
- Taiwan (5):
  - Taichung Veterans General Hospital ( Site 3703), Taichung
  - National Cheng Kung University Hospital ( Site 3702), Tainan
  - National Taiwan University Hospital ( Site 3701), Taipei
  - Mackay Memorial Hospital ( Site 3704), Taipei
  - Linkou Chang Gung Memorial Hospital ( Site 3705), Taoyuan District
- Thailand (4):
  - Ramathibodi Hospital. ( Site 3802), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 3801), Bangkok, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 3804), Chiang Mai
  - Faculty of Medicine - Khon Kaen University ( Site 3803), Khon Kaen
- United Kingdom (10):
  - University Hospitals Sussex NHS Foundation Trust ( Site 4011), East Sussex, Brighton And Hove
  - Addenbrookes Hospital ( Site 4002), Cambridge, Cambridgeshire
  - University College London Hospital ( Site 4001), London, London, City of
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 4006), London, London, City of
  - Hammersmith Hospital ( Site 4010), London, London, City of
  - Western General Hospital ( Site 4012), Edinburgh, Midlothian
  - Royal Marsden Hospital (Sutton) ( Site 4005), London, Surrey
  - Leicester Royal Infirmary ( Site 4008), Leicester
  - Maidstone Hospital ( Site 4007), Maidstone
  - The Christie NHS Foundation Trust ( Site 4003), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/